CLINICAL TRIAL: NCT07332364
Title: Additional Effects of Sensory Integration Along With Focused Regimen Exercises on Kinaesthesia & Proprioception in Diabetic Peripheral Neuropathy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2025/15
Record Dates: First submitted 2025-12-30; First posted 2026-01-12 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Diabetic Neuropathy; Proprioception
Keywords: physical therapy; diabetic neuropathy; kinesthesia; proprioception; exercises
MeSH Terms: conditions — Diabetic Neuropathies; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sensory integration exercises along with focused regimen exercise (Experimental): 8-week progressive balance, strength, and sensory stimulation program, performed three sessions per week. Weeks 1-2 focused on sensory activation and basic strengthening, including textured ball rolling and brushing of the feet, ankle circles, toe scrunches, double-leg calf raises, resistance-band ankle exercises, weight-shifting on a foam pad, and 10 minutes of TENS at comfortable intensity. Weeks 3-4 progressed to single-leg calf raises, tandem walking, balance board training, and reduced TENS duration (8 minutes). Weeks 5-6 emphasized dynamic balance and functional strength through single-leg balance with ball toss, barefoot walking on uneven surfaces, squats, multidirectional stepping, and 6 minutes of TENS. Weeks 7-8 advanced balance challenges with obstacle walking, wobble board training with minimal support, barefoot balance with ball toss on uneven ground, weighted calf raises, single-leg stance, and eyes-closed balance exercises to enhance proprioception and postural control.
  Interventions: Procedure: Sensory integration and focused regimen
- focused regimen exercises (Active Comparator): The exercise program was delivered over 8 weeks, with participants completing three sessions per week and progressing in difficulty. During weeks 1-2, the focus was on basic strengthening and ankle control through double-leg calf raises and resistance-band ankle exercises, including dorsiflexion, plantarflexion, inversion, and eversion to improve ankle mobility and muscle activation. Weeks 3-4 introduced unilateral strengthening and functional balance tasks, such as single-leg calf raises, step-ups using a low platform, and balance board training to enhance postural stability. In weeks 5-6, the program emphasized functional lower-limb strength and dynamic balance using double-leg squats and multidirectional stepping exercises. During weeks 7-8, the intensity was increased with weighted calf raises, prolonged single-leg stance exercises, and eyes-closed balance training to challenge proprioception and postural control.
  Interventions: Procedure: Focused Regimen Exercise

INTERVENTIONS:
Procedure: Sensory integration and focused regimen — 3 sessions/week 1-2 weeks : textured ball and brush on feet. (3-5 min/foot). Ankle circles, toe scrunches.10 reps x 2 sets, Tens 10min, 2 sets calf raises (10 reps). resistance band (10 reps x 2 sets). 3-4 weeks: Shift weight side-to-side and forward-backward on foam pad (10 reps x 2 sets). calf raises, progressing to single-leg calf raises 10 reps x 2 sets. Step-ups: Step up and down 10 reps x 2 sets. Standing on board 30 sec. Open. 5-6 weeks: Tandem walking. Tens 8min. Balance on one leg while catching a ball (20-30 sec). barefoot walking (grass, gravel).Tens 6min. Double-leg squats10 reps x 1 set. side-to-side and forward-backward stepping 10 reps x 2 sets. 7-8 weeks: Walk over & around obstacles. Balance wobble board for 30 sec-2 reps. Balance barefoot on uneven terrain while catching a ball. Weighted calf raises 10 reps x 3 sets. Standing on firm surface for 30 sec. Eyes close, Single-leg stance 10 reps x 3 sets
  Arms: sensory integration exercises along with focused regimen exercise
Procedure: Focused Regimen Exercise — 3 sessions/week 1-2 weeks Perform 2 sets of calf raises (10 reps). Use a resistance band (green colour) 10 reps x 2 sets. 3-4 weeks: calf raises, progressing to single-leg calf raises. 10 reps x 2 sets Step-ups: Step up and down on a low step 10 reps x 2 sets. Standing on board for 30 sec. Open. 5-6 weeks :Double-leg squats10 reps x 1 set. Perform side-to-side and forward-backward stepping 10 reps x 2 sets Weighted . 7-8 weeks: calf raises 10 reps x 3 sets. Standing on firm surface for 30 sec. Eyes close, Single-leg stance on firm ground10 reps x 3 sets
  Arms: focused regimen exercises

SUMMARY:
This study aims to evaluate Additional Effects of sensory integration along with focused regimen exercises on kinaesthesia & proprioception in Diabetic peripheral neuropathy Peripheral neuropathy a Condition occur when the nerves outside the brain and spinal cord are damaged. It affects the upper and lower extremity. The estimated prevalence of peripheral neuropathy in patients with diabetes in Pakistan is around 43%. The condition is more common in those who have poorly controlled diabetes. Signs and symptoms include Numbness, tingling, Pain, which may be burning, stabbing or shooting, unusual touch-based sensations (dysesthesia), Muscle weakness, Total or partial loss of sensation in feet, like not feeling pain from foot injuries, loss of position and movement sense.

Kinaesthesia and proprioception are defined as awareness of the position and movement of the body parts by sensory organs (proprioceptors) in the muscles and joints. Uncoordinated movement, clumsiness, poor postural control are common symptoms. Multiple treatment options are available for training kinaesthesia and proprioception impairments in peripheral neuropathy including use of electrotherapeutic agents, proprioception exercises, sensory integration, and focused regimen exercises. Current study will be RCT on 40 participants recruited on the basis of inclusion criteria which are Diagnosed as Type 2 Diabetic peripheral neuropathy (DPN) by physician in the age group of 45-65 Years in Both genders with type 2 Diabetes. Patients with moderate neuropathy according to Michigan nephropathy screening tool and having the ability to walk with or without assistance. Participants will be randomly and equally divided into two groups; group A will be receiving focused regimen exercises and group B will be receiving both sensory integration exercises along with focused regimen exercises.

The treatment will be given for 45min, 3 days a week for total of 8 weeks. The assessment will be conducted at baseline by (Michigan neuropathy screening tool, Brief kinaesthesia test (BKT), Modified Clinical Test of Sensory Interaction for balance (mCTSIB), Norfolk quality of life for diabetic neuropathy), and final assessment will be conducted after 8 weeks of treatment.

DETAILED DESCRIPTION:
Peripheral neuropathy a Condition occurs when the nerves outside the brain and spinal cord are damaged. It affects the upper and lower extremity. The estimated prevalence of peripheral neuropathy in patients with diabetes in Pakistan is around 43%. The condition is more common in those who have poorly controlled diabetes. Signs and symptoms include Numbness, tingling, Pain, which may be burning, stabbing or shooting, unusual touch-based sensations (dysesthesia), Muscle weakness, Total or partial loss of sensation in feet, like not feeling pain from foot injuries, loss of position and movement sense. Although there are many possible causes of peripheral neuropathy, the most prevalent subtype, diabetic peripheral neuropathy (DPN), can lead to significant complications ranging from paresthesia to loss of limb and life. Early assessment of symptoms of peripheral polyneuropathy helps avoid neuropathic foot ulcers to combat potential morbidity and mortality resulting from the pathophysiologic poor wound healing potential, which can lead to limb compromise, local to systemic infection, septicemia, and even death. Early peripheral neuropathy may present as sensory alterations that are often progressive, including sensory loss, numbness, pain, or burning sensations in a "stocking and glove" distribution of the extremities. Later stages may involve proximal numbness, distal weakness, or atrophy. Early peripheral neuropathy may present as sensory alterations that are often progressive, including sensory loss, numbness, pain, or burning sensations in a "stocking and glove" distribution of the extremities. Later stages may involve proximal numbness, distal weakness, or atrophy. kinesthetic sensation or joint sensation and movement of limbs has been a subject of surmise for more than 400 years. It is defined as awareness of the position and movement of the parts of the body by means of sensory organs (proprioceptors) in the muscles and joints. It is a function through which the investigators can tell where our body parts are located even when our eyes are closed or when the investigators are not looking at our body. It is basically controlled by muscle spindles, joint and skin receptors. According to the hypothesis by Yin4 , basal ganglia control the speed of movement through kinesthetic re-afferent input. The entire nervous system is responsible for kinesthetic sense. kinesthesia is important component in muscle memory and coordination. Burning and stabbing pain in the feet and lower limbs can have a significant impact on the activities of daily living, including walking, climbing stairs and sleeping. Peripheral neuropathy in particular is often misdiagnosed or under-diagnosed because of a lack of awareness among both patients and physicians. The underestimation of peripheral neuropathy is highly prevalent in the South-East Asia region due to a lack of consensus guidance on routine screening and diagnostic pathways. Joint position sense is important to maintain stability. Rehabilitation of impaired kinesthesia includes use of different textures, shapes, weight in order to assist sensory reeducation. To integrate proprioception balance training is used. Repetitive practice of stimulation is frequently practiced. In physiotherapy management the investigators mostly concentrate on neuropathic pain, weakness but neglect proprioceptive problems. Identifying them and treating at right time is very important to avoid progression as well as complications of the disease. Sensory nerves carry important proprioceptive information about the position of our body parts in relation to each other and to the surrounding environment. Proprioceptive signals are derived from mechanoreceptors located in the skin, joints, tendons, ligaments, and muscles. In particular, muscle spindles play a major role in the sense of proprioception throughout the range of joint motion. Collectively, the action potentials generated from the mechanoreceptors are carried through afferent nerve fibers and processed in the central nervous system (CNS) to provide the sense of proprioception. Proprioceptive disorders may occur when thick fibers are affected in diabetic neuropathy. This can lead to impaired joint stabilization and increased risk of falls and fractures. Loss of foot-sole input goes along with large-fiber dysfunction in intrinsic foot muscles. Diabetic patients have an elevated risk of falling, and vision and vestibular compensation strategies may be inadequate. The investigators touch on the effects of nerve stimulation onto cortical and spinal excitability, which may participate in plasticity processes, and on exercise interventions to reduce the impact of neuropathy. Even if the short-term effect of a sensory volley produced by electrical stimulation of a peripheral nerve (either cutaneous or muscular261) reaching the sensory motor cortex is far beyond the scope of this short article, the investigators would like to remind that this mere direct input plays a remarkable role in modifying the cortical excitability. These effects (e.g., short-latency afferent inhibition, afferent facilitation, and long-latency afferent inhibition) have been attributed a role in cortical plasticity. A large number of mechanoreceptors and sensory fibers are recruited when stimulated by TENS at various frequencies, intensities and durations. Proprioceptors being specialized mechanoreceptors relay continuous detailed knowledge about the positions of the various body parts to the cortex, aiding in their spatial position. High frequency TENS when applied to the lower limb had a positive influence over the postural sway in a study done by Dickstein et al. They concluded that electrical stimulations decrease the mechanoreceptor thresholds and thus improve proprioception. studies suggest that there is postural instability in people with DPN which increases with age and duration of diabetes. Multidirectional postural sway was observed in most of the studies with medio-lateral instability encountered in more cases. Significant improvement in timed up and go test, single leg stance test, Berg balance scale, and other outcome measures post physiotherapy intervention were reported. Literature suggests that multidirectional postural instability is present in DPN patients.

ELIGIBILITY:
Inclusion Criteria:

* Participants Diagnosed as Type 2 DPN by physician.
* Age between 45-65 Years.
* Both genders males and females.
* Patient with moderate neuropathy according to Michigan neuropathy screening tool.
* Ability to walk with or without assistance

Exclusion Criteria:

* Unstable Cardiovascular diseases. (Myocardial infarction, Heart failure, Coronary artery disease, Arrythmias)
* Severe visual disorders. (Cataracts, Glaucoma, Macular degeneration)
* Severe musculoskeletal problems of lower limb (Fractures).
* Any metal implant. (presence of pacemaker, artificial joints or screws in lower extremity).
* Unable to follow basic instructions

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-09-15 (Actual); Primary Completion 2025-10-26 (Actual); Study Completion 2025-12-20 (Actual)

PRIMARY OUTCOMES:
Kinesthesia and Proprioception | 8 weeks
  The Brief kinaesthesia Test (BKT) is used to assess kinaesthesia and proprioception in the ankle by evaluating joint position sense (JPS) and movement detection (Threshold to Detect Passive Motion - TTDPM).
  Scoring Interpretation of JPS:
  0-2 error = Good proprioception 2.1-4 error= mild impairment 4.1-7 error = Moderate impairment >7 error = Poor proprioception Movement Detection Test (Threshold to Detect Passive Motion - TTDPM) Determine the smallest movement the participant can detect.
  Scoring Interpretation of TTDPM:
  0-2 threshold = Excellent proprioception 2.1-4 threshold = Mild impairment 4.1-6 threshold= moderate impairment >6.0 threshold = Poor proprioception
Quality of Life of Diabetic Peripheral Neuropathy Patients | 8 weeks
  The Norfolk QoL-DN is a validated questionnaire used to assess the impact of diabetic neuropathy (DN) on a patient's quality of life. It covers sensory, autonomic, motor, and psychosocial aspects of neuropathy.
  Minimum score = 0 (No neuropathy) Maximum score = 140 (Severe neuropathy impact) Interpretation Total Score Range Severity 0-20 No neuropathy 21-40 Mild neuropathy 41-70 Moderate neuropathy >70 Severe neuropathy A higher score indicates worse neuropathic impact.
Sensory Balance | 8 weeks
  The Modified Clinical Test of Sensory Interaction in Balance (mCTSIB) evaluates postural control by testing balance under different sensory conditions. It is used to assess impairments in vestibular, somatosensory, and visual systems, making it valuable for diagnosing balance disorders.
  Maximum Score = 120 seconds (if all conditions are completed successfully). Minimum Score = 0 seconds (if unable to balance in any condition). Scoring Interpretation Total Score (out of 120 sec) Balance Impairment Level >110 sec Normal Balance 90-109 sec Mild Impairment 60-89 sec Moderate Impairment <60 sec Severe Impairment

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Islamabad, Pakistan